CLINICAL TRIAL: NCT03854188
Title: Acupuncture for Relieving Chronic Pelvic Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principle investigator is leaving institution.
Sponsor: William Xu, MD (Other)
Responsible Party: Sponsor-Investigator, William Xu, MD, Associate Anesthesiologist, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201808791
Record Dates: First submitted 2019-02-05; First posted 2019-02-26 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Pelvic Pain
Keywords: acupuncture
MeSH Terms: conditions — Pelvic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture treatment (Experimental): Patients diagnosed with chronic pelvic pain will be offered acupuncture treatment as an adjuvant therapy to standard of care treatment.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Use acupuncture therapy in the treatment of chronic pelvic pain.

SUMMARY:
Individuals with chronic pelvic pain will be identified, consented and enrolled in this study in which acupuncture will be offered in addition to current standards of care. The primary outcome will assess if there is a reduction of pain intensity from the baseline to 6 months as a result of treatment.

DETAILED DESCRIPTION:
Chronic pelvic pain as defined by the American College of Obstetricians and Gynecologists is "noncyclic pain of 6 or more months duration that localizes to the anatomic pelvis, anterior abdominal wall at or below the umbilicus, the lumbosacral back or the buttocks and is of sufficient severity to cause functional disability or lead to medical care". This has devastating consequences both monetarily as well as emotionally and can lead to opioid addiction, depression and even suicide.

Acupuncture has been used to treat pain in China for millenniums and was one of the more effective ways to treat pain before morphine was discovered. Acupuncture is feasible, economic and a safe way to treat chronic pain.

Patients with chronic pelvic pain will be identified and offered participation in the study. After the consent process is completed, patients will undergo a brief physical exam to rule out acute symptoms. The patient will be asked to complete a baseline pain inventory and genitourinary pain index survey before proceeding with acupuncture treatment. Qualified patients will be requested to accept acupuncture treatments twice weekly for 12 consecutive weeks. Each week the patient will be asked to report their current medications and changes in the dosage as well as their narcotic (opioid) doses and any changes in the dosages. Patients will be followed up monthly for up to 3 months after treatment completion by phone to record their pain inventory as well as their genitourinary pain index survey.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pelvic pain persisting for at least 6 months
* English speaking
* Able to provide informed consent

Exclusion Criteria:

* Unable to provide informed consent
* Pregnant
* Prisoners
* Morbid obesity (BMI >40, or > 36 associated with hypertension and diabetes)
* Severe cardiac disease
* Active chemotherapy or radiation therapy
* Skin infections or lesions
* Severe COPD
* Neuropathy
* Previous stroke
* Paralysis
* Needle phobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure pelvic specific pain | Three months
  Subjects will report baseline pain scores using the Genitourinary Pain Index (GUPI). The index is used to quantify the severity of pelvic pain experienced by the patient. It is a self-reporting condition specific questionnaire (gender specific) that is scored based on information provided by the patient. The scale is 0 to 5 with 0 indicating never experienced and 5 indicating being always present. The same index will be used at the end of treatment to determine the post-treatment scores and compared to baseline scores.
Measure generalized body pain | Three months
  Subjects will report initial baseline pain scores using the Brief Pain Inventory (BPI). The BPI assesses the severity of pain experienced by the patient and calculates pain's impact on daily functioning. It is self-reported and uses a numerical scale where 0 indicates no pain and 10 indicating pain as bad as the patient can image. The patient will report again using the BPI at the end of treatment and the values obtained will be compared to the baseline scores.

SECONDARY OUTCOMES:
Measure pain score after treatment-1 month (GUPI) | One month post treatment
  Subjects reported baseline pain scores using the Genitourinary Pain Index (GUPI). The index is used to quantify the severity of pelvic pain experienced by the patient. It is a self-reporting condition specific questionnaire (gender specific) that is scored based on information provided by the patient. The scale is 0 to 5 with 0 indicating never experienced and 5 indicating being always present. The same index will be used 1 month following the end of treatment and compared to baseline scores.
Measure pain score after treatment-1 month (BPI) | One month post treatment
  Subjects reported baseline pain scores using the Brief Pain Inventory (BPI). The BPI assesses the severity of pain experienced by the patient and calculates pain's impact on daily functioning. It is self-reported and uses a numerical scale where 0 indicates no pain and 10 indicating pain as bad as the patient can image. The BPI will be used 1 month following the end of treatment and compared to baseline scores.
Measure pain score after treatment-2 months (GUPI) | Two months post treatment
  Subjects reported baseline pain scores using the Genitourinary Pain Index (GUPI). The index is used to quantify the severity of pelvic pain experienced by the patient. It is a self-reporting condition specific questionnaire (gender specific) that is scored based on information provided by the patient. The scale is 0 to 5 with 0 indicating never experienced and 5 indicating being always present. The same index will be used 2 months following the end of treatment and compared to baseline scores.
Measure pain score after treatment-2 months (BPI) | Two months post treatment
  Subjects reported baseline pain scores using the Brief Pain Inventory (BPI). The BPI assesses the severity of pain experienced by the patient and calculates pain's impact on daily functioning. It is self-reported and uses a numerical scale where 0 indicates no pain and 10 indicating pain as bad as the patient can image. The BPI will be used 2 months following the end of treatment and compared to baseline scores.
Measure pain score after treatment-3 months (GUPI) | Three months post treatment
  Subjects reported baseline pain scores using the Genitourinary Pain Index (GUPI). The index is used to quantify the severity of pelvic pain experienced by the patient. It is a self-reporting condition specific questionnaire (gender specific) that is scored based on information provided by the patient. The scale is 0 to 5 with 0 indicating never experienced and 5 indicating being always present. The same index will be used 3 months following the end of treatment and compared to baseline scores.
Measure pain score after treatment-3 months (BPI) | Three months post treatment
  Subjects reported baseline pain scores using the Brief Pain Inventory (BPI). The BPI assesses the severity of pain experienced by the patient and calculates pain's impact on daily functioning. It is self-reported and uses a numerical scale where 0 indicates no pain and 10 indicating pain as bad as the patient can image. The BPI will be used 2 months following the end of treatment and compared to baseline scores.

CONTACTS AND LOCATIONS:
Overall Officials: William Xu, MD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data (IPD) collected during the trial, after deidentification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: IPD will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal

REFERENCES:
- [Background] ACOG Committee on Practice Bulletins--Gynecology. ACOG Practice Bulletin No. 51. Chronic pelvic pain. Obstet Gynecol. 2004 Mar;103(3):589-605. No abstract available. PMID 14990428
- [Background] Mathias SD, Kuppermann M, Liberman RF, Lipschutz RC, Steege JF. Chronic pelvic pain: prevalence, health-related quality of life, and economic correlates. Obstet Gynecol. 1996 Mar;87(3):321-7. doi: 10.1016/0029-7844(95)00458-0. PMID 8598948
- [Background] Zhang R, Lao L, Ren K, Berman BM. Mechanisms of acupuncture-electroacupuncture on persistent pain. Anesthesiology. 2014 Feb;120(2):482-503. doi: 10.1097/ALN.0000000000000101. PMID 24322588
- [Background] MacPherson H, Vertosick EA, Foster NE, Lewith G, Linde K, Sherman KJ, Witt CM, Vickers AJ; Acupuncture Trialists' Collaboration. The persistence of the effects of acupuncture after a course of treatment: a meta-analysis of patients with chronic pain. Pain. 2017 May;158(5):784-793. doi: 10.1097/j.pain.0000000000000747. PMID 27764035
- [Background] Vickers AJ, Vertosick EA, Lewith G, MacPherson H, Foster NE, Sherman KJ, Irnich D, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for Chronic Pain: Update of an Individual Patient Data Meta-Analysis. J Pain. 2018 May;19(5):455-474. doi: 10.1016/j.jpain.2017.11.005. Epub 2017 Dec 2. PMID 29198932
- [Background] Ernst, E., White A. Acupuncture - A Scientific Appraisal. ISBN#978-0-7506-4163-0